CLINICAL TRIAL: NCT03318237
Title: Ultra High Field MRI of Focal Pediatric Epilepsy
Status: Terminated | Type: Observational
Why Stopped: PI moved to a different institution.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00125321
Record Dates: First submitted 2017-10-06; First posted 2017-10-23 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with focal epilepsy: Patients undergoing ultra high field MRI of the brain

SUMMARY:
Epilepsy affects a significant number of children in the United States. The majority of patients achieve control of their seizures by conventional treatment strategies including medications. However, one third of patients do not achieve satisfactory seizure control with medications alone. Ketogenic diet and lifestyle modifications may also be tried. In some of these children, the seizure focus can be localized to one area of the brain and the seizures are resistant to conservative treatment strategies. These children may have subtle structural/developmental abnormalities in their brain, the most frequent of which is focal cortical dysplasia. These are localized areas of abnormal lamination of the cerebral cortex that can be extremely subtle and difficult to detect, even with state of the art magnetic resonance imaging (MRI). More importantly, these lesions may be amenable to surgical resection resulting in marked decrease in frequency or even resolution of seizures.

MRI is a noninvasive imaging modality without ionizing radiation that has played a central role in the assessment of anatomy, physiology/pathophysiology of children with epilepsy. It is particularly useful in children with refractory focal epilepsy. Prior studies have shown that high resolution, high-field (3T) MR imaging of the brain helps to identify subtle focal epileptogenic abnormalities, including focal cortical dysplasia, in some patients. However, there is scarce data directly comparing the performance of ultra high-field (7T) MRI, currently an investigative technique offering optimized contrast and signal-to-noise rations and superior spatial resolution, with clinically available 3T MR imaging.

The purpose of this study is to evaluate whether ultra high-field (7T) MR imaging improves detection and characterization of subtle structural epileptogenic abnormalities in children with focal epilepsy.

The importance of this research is that identification of a focal epileptogenic lesion in children with refractory epilepsy has fundamental management implications, as surgical removal of such lesion may dramatically improve outcomes and the chance of seizure freedom.

DETAILED DESCRIPTION:
1. Abstract Epilepsy affects a significant number of children in the United States. The majority of patients achieve control of their seizures by conventional treatment strategies including medications. However, one third of patients do not achieve satisfactory seizure control with medications alone. Ketogenic diet and lifestyle modifications may also be tried. In some of these children, the seizure focus can be localized to one area of the brain and the seizures are resistant to conservative treatment strategies. These children may have subtle structural/developmental abnormalities in their brain, the most frequent of which is focal cortical dysplasia. These are localized areas of abnormal lamination of the cerebral cortex that can be extremely subtle and difficult to detect, even with state of the art magnetic resonance imaging (MRI). More importantly, these lesions may be amenable to surgical resection resulting in marked decrease in frequency or even resolution of seizures.

   MRI is a noninvasive imaging modality without ionizing radiation that has played a central role in the assessment of anatomy, physiology/pathophysiology of children with epilepsy. It is particularly useful in children with refractory focal epilepsy. Prior studies have shown that high resolution, high-field (3T) MR imaging of the brain helps to identify subtle focal epileptogenic abnormalities, including focal cortical dysplasia, in some patients. However, there is scarce data directly comparing the performance of ultra high-field (7T) MRI, currently an investigative technique offering optimized contrast and signal-to-noise rations and superior spatial resolution, with clinically available 3T MR imaging.

   The purpose of this study is to evaluate whether ultra high-field (7T) MR imaging improves detection and characterization of subtle structural epileptogenic abnormalities in children with focal epilepsy.

   The importance of this research is that identification of a focal epileptogenic lesion in children with refractory epilepsy has fundamental management implications, as surgical removal of such lesion may dramatically improve outcomes and the chance of seizure freedom.
2. Objectives (include all primary and secondary objectives)

   The objectives of Investigators' project are:

   To evaluate the performance of 7T MRI in detecting structural abnormalities in children who have had 3T MRI-negative focal epilepsy.

   To characterize conventional and advanced neuroimaging features of epileptogenic lesions such as cortical dysplasias and neuroglial tumors at 7T MRI.
3. Background High-resolution brain MRI is currently an integral component in the diagnostic evaluation of children with focal epilepsy. When focal epileptogenic abnormalities are identified, such as cortical dysplasia, the management strategy includes evaluation for potential surgical resection, which may dramatically improve outcome. The current clinical state of the art of 3T MRI has superior sensitivity over conventional 1.5T MRI. However focal cortical dysplasia remains one of the most common pathological diagnoses after pediatric epilepsy surgery, even when not detected by current MRI exams.
4. Study Procedures

   1. Study design, including the sequence and timing of study procedures. The investigators plan to perform 7T brain MRI in children with the diagnosis of epilepsy and findings on EEG suggestive of a focal structural abnormality. The 7T MRI exams will be performed at Kennedy Krieger Institute (KKI) as part of their outpatient evaluation. The investigators plan to accrue approximately 50 participants.

      Before recruiting children with epilepsy, approximately 2-10 healthy adult volunteers will be recruited for the purpose of optimizing the imaging acquisition protocol. These adults will be consented using a separate consent form, also attached to this application.

      Children will be eligible if they have already had a 3T MRI examination and do not have any contraindications to MR examinations. A consent form signed by the patients' parent/legal care giver will be required to indicate agreement to participate in the study. In addition, a consent form signed by the patient (if over 15 year of age) or an assent form signed by the patient (if between 8-15 years of age) will be required to indicate agreement to participate. Patient charts will be reviewed for history and diagnosis.
   2. Study duration and number of study visits required of research participants. The anticipated duration of this study will be 2-5 years beginning in April 2017. The 7T MRI exam will be performed in a single visit. This project may involve one additional trip to the hospital for patient subjects.
   3. Blinding, including justification for blinding or not blinding the trial, if applicable.

      N/A
   4. Justification of why participants will not receive routine care or will have current therapy stopped.

      N/A
   5. Justification for inclusion of a placebo or non-treatment group. N/A
   6. Definition of treatment failure or participant removal criteria. Removal criteria will be defined as participants who are unable to tolerate the MR procedure due to previously unknown claustrophobia, inability to tolerate lying still for the exam period, or due to presence of ferromagnetic implants preventing imaging.
   7. Description of what happens to participants receiving therapy when study ends or if a participant's participation in the study ends prematurely.

Not applicable. This is not a treatment study.

Data collection and management will be implemented with the following guidelines to ensure their confidentiality and safety:

1. Confidentiality of Data: A master list separate from data forms that have only a study number will be used to maintain confidentiality of data.
2. Security: The master list and backup copy will both be kept only on secure Johns Hopkins computers. Only de-identified data will be stored on a non-Johns Hopkins personal computer.
3. Anonymization: The identifiers will be destroyed after publication. The other data will be retained for three years.
4. Confidentiality: All data and records generated during this study will be kept confidential in accordance with Institutional policies and HIPAA on subject privacy and that the Investigator and other site personnel will not use such data and records for any purpose other than conducting the study. Safeguards are described under Data Collection and Management.
5. Inclusion/Exclusion Criteria

   a. Inclusion Criteria i. Male or female children between 6-21 years of age undergoing an MRI for focal epilepsy at the Johns Hopkins Hospital OR ii. Adult healthy volunteer. iii. Willing to undergo an additional MRI exam in the 7T scanner at Kennedy Krieger Institute.

   b. Exclusion Criteria i. Presence of any contraindication to MR examinations as defined by MRI Safety Screening Sheet ii. History of Metal in the Skull/Eyes iii. Pregnancy at the time of the scan iv. Patient subjects in unstable clinical condition
6. Drugs/ Substances/ Devices

   1. The rationale for choosing the drug and dose or for choosing the device to be used.

      Only patients with a clinical indication for brain MRI examination will undergo 7T MRI. All examinations will be performed without intravenous contrast and in an outpatient setting, without the need for deep sedation or general anesthesia. Although classified by FDA as an investigational device, the 7T MR system has been ruled as a non-significant risk device by the same agency. This finding is stipulated in Guidance for Industry and FDA Staff --Criteria for Significant Risk Investigations of Magnetic Resonance Diagnostic Devices issued July 14, 2003. A copy of the ruling has been uploaded in Section 3.0 for your review. In well over 1000 studies done at 7T in the last decade at multiple institutions (University of Minnesota, Massachusetts General Hospital, NIH), no significant risks have been found. Some subjects have experienced dizziness. A potential concern with MR studies at high fields is radiofrequency heating due to radiofrequency power deposition in the subject. The FDA has set strict guidelines to guard against this risk. Such power deposition increases with the square of the magnetic field strength. However, even at 7T it is possible to stay well within these guidelines, especially with the pulse sequences the investigators will employ. To be 100% sure of compliance with FDA guidelines, the software of the manufacturer monitors power deposition continuously and scans are not possible to implement if the power deposition would exceed guidelines.

      Documents have been uploaded in Section 3.0 regarding federal guidelines supporting the position that a 7 Tesla MR scanner represents no significant risk to human subjects.

      Theoretical concepts and prior clinical studies justify the interest in applying high-resolution, ultra high-field MRI as a tool to evaluate detailed brain anatomy and physiology in children with focal epilepsy. Most studies comparing the diagnostic yield of 3T versus 1.5T imaging in detecting structural lesions in patients with focal epilepsy reached positive conclusions concerning the rates of newly detected lesions at 3T Very few comparative studies have investigated the diagnostic yield of 7T with respect to conventional MRI, however these included both examinations performed at 1.5T and at 3T.

      The employment of 7T MRI provides superior capability in characterizing anatomical and physiological brain parameters. In collaboration with MR physicists affiliated with Johns Hopkins and with Kennedy Krieger Institute, our imaging acquisition protocol should include:
      * High-resolution anatomical sequences, such as volumetric T1-weighted MP2RAGE and 2D gray-white tissue border enhancement (TBE) Fast Spin Echo (FSE)-Inversion Recovery (IR). These images are optimal for evaluating the interface between the cortex and the juxtacortical white matter when attempting to detect subtle focal cortical dysplasias, an important cause of focal refractory epilepsy in children.
      * Susceptibility-weighted imaging. 7T has been shown to offer superior sensitivity in detecting abnormal blood products and iron deposition in the cerebral parenchyma, in addition to the exquisite depiction of the normal and abnormal cerebral venous anomaly. These images may also be used for subjective evaluation of oxygen extraction fraction in the brain, and for quantitative mapping of iron deposition.
      * Diffusion tensor imaging (DTI) and diffusion kurtosis imaging (DKI). Both techniques explore the diffusivity of water molecules in the intra- and extracellular spaces of the brain, along with the directionality of movement. The acquisition generates parameters of white matter integrity and anisotropy, including mean diffusivity, longitudinal and radial diffusivity, and fractional anisotropy. With this information, detailed in vivo maps of white matter fibers (tractography) can be produced, as well as maps of anatomic connectivity (connectome). DKI is a novel diffusion imaging technique that explores the non-Gaussian distribution of white matter molecules and is able to further characterize the complexity of white matter microstructure. DKI has thus far been scarcely explored in the study of pediatric neurological disorders.
      * Resting-state functional MRI. Several studies have shown disturbance of functional pathways in children with focal refractory epilepsy. This technique relies on the blood-oxygen level dependent (BOLD) effect, does not require tasks as in other Functional MRI (fMRI) acquisitions, and can be postprocessed to generate maps of functional connectivity.
      * MR Spectroscopy (MRS): 1H MRS is a noninvasive imaging technique that can easily be added to the conventional MRI sequences and is able to measure metabolism in the brain. Metabolic changes arising from pathology that can be visualized by MRS may not be apparent from anatomy. During a seizure, the metabolic demands exceed the supply of oxygen and nutrients to the portion of the brain that is undergoing the enhanced electric activity. Under these circumstances, metabolic changes can be detected by MRS, including the production of lactate and, if prolonged, the reduction of N-Acetyl Aspartate (NAA), and an increase in Cho. These abnormalities can still be observed after seizure activity ceases. Another common clinical scenario for the use of MRS is temporal-lobe epilepsy (TLE) to help localize the source of the seizures.

      Images acquired from 7T MRI examinations will not be used in isolation to guide patient care. In the event that 7T discloses a focal structural abnormality of the brain that was not detected at 3T MRI, this finding will be evaluated by a multidisciplinary team responsible for care of the particular patient. Management decisions will then be suggested to the patient and family considering all the clinical, electrographic, and neuroimaging data available.
   2. Justification and safety information if FDA approved drugs will be administered for non-FDA approved indications or if doses or routes of administration or participant populations are changed.

      Not applicable.
   3. Justification and safety information if non-FDA approved drugs without an Investigational New Drug (IND) will be administered.

   Not applicable.
7. Study Statistics

   1. Primary outcome variable. The primary outcome variable is the sensitivity of 7T brain MRI in the detection of subtle cortical abnormalities in children with focal epilepsy.
   2. Secondary outcome variables. The secondary outcome variables include subjective characterization of subtle epileptogenic lesions, and quantitative metrics from advanced MR sequences such as apparent diffusion coefficient (ADC) and fractional anisotropy (FA) may be obtained from DTI sequences. Quantitative parameters may also be obtained from other imaging techniques such as MR spectroscopy.
   3. Statistical plan including sample size justification and interim data analysis. N/A
   4. Early stopping rules. N/A
8. Risks

   1. Medical risks, listing all procedures, their major and minor risks and expected frequency.

      All participants will undergo the informed consent process. Children over the age of 15 will be asked to document their consent by signing the consent form. Children between the ages of 8 and 15 years of age will be asked to indicate their assent by signing the assent document. Assent will be obtained for children <8 years of age by monitoring visual and vocal indications as well as body language. Parents of all children will be asked to document their consent of the procedure on the consent form.

      The effects of magnetic fields in an MRI scanner have been extensively studied, and there are no known risks with an MRI exam. Participants may, however, be bothered by feelings of confinement (claustrophobia), and by the noise made by the image acquisition during the procedure.
   2. Steps taken to minimize the risks. Participants will be asked about contraindications to MR examinations (as outlined by the MRI screening sheet). Participants will wear earplugs and earphones while in the magnet. Participants may not participate in this study if they have a pacemaker, an implanted defibrillator or other implanted electronic or metallic devices.
   3. Plan for reporting unanticipated problems or study deviations. Adverse events, unanticipated problems, and study deviations will be reported to the IRB in writing by study personnel within 5 days of learning of the event. Serious adverse events will be reported immediately.
   4. Legal risks such as the risks that would be associated with breach of confidentiality.

      There are no known or anticipated legal risks associated with participating in this study.
   5. Financial risks to the participants. There are no known or anticipated financial risks associated with participating in this study.
9. Benefits

   a. Description of the probable benefits for the participant and for society. i. Individual participant

   Individual participants may benefit by receiving higher end, non-invasive, non-contrast MR imaging studies that may (or may not) increase sensitivity and specificity of diagnosis and prognosis.

   ii. Society Society may benefit if investigators are able to establish the value of 7T MR imaging in focal pediatric epilepsy. By developing a high-resolution 7T brain MRI protocol for pediatric epilepsy, the data obtained from these exams may serve as the basis to alter diagnostic workup. This may ultimately improve early detection and characterization of lesions, and guide surgical planning, and may facilitate better outcomes.
10. Payment and Remuneration

    a. Detail compensation for participants including possible total compensation, proposed bonus, and any proposed reductions or penalties for not completing the protocol.

    All studies will be performed in addition to a clinically indicated MRI appointment. No additional costs or billing will be generated to the patients. Subjects may receive a copy of their images on compact disc upon request.
11. Costs a. Detail costs of study procedure(s) or drug (s) or substance(s) to participants and identify who will pay for them.

Patient subjects will not incur any additional costs directly related to their participation in this project. The 7T MRI exams will be funded by a research grant.

ELIGIBILITY:
Inclusion Criteria:

* Male or female children between 6-21 years of age undergoing an MRI for focal epilepsy at the Johns Hopkins Hospital OR ii. Adult healthy volunteer. iii. Willing to undergo an additional MRI exam in the 7T scanner at Kennedy Krieger Institute.

Exclusion Criteria:

* Presence of any contraindication to MR examinations as defined by MRI Safety Screening Sheet ii. History of Metal in the Skull/Eyes iii. Pregnancy at the time of the scan iv. Patient subjects in unstable clinical condition

Ages: 6 Years to 21 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children with the diagnosis of epilepsy and findings on EEG suggestive of a focal structural abnormality.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Detection rate of subtle structural epileptogenic abnormalities in children with focal epilepsy. | At the time of brain MRI exam.
  The rate of abnormal findings detected by 7T MRI in children with focal epilepsy will be recorded, as well as their location and relationship with abnormal electroencephalographic (EEG) findings. These findings include areas of malformation or scarring (dysplasia or gliosis) in the cerebral cortex, for example.

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States